CLINICAL TRIAL: NCT02266368
Title: A Randomized Controlled Trial Comparing Antimicrobial Coated (Silver Sulfadiazine) Ureteral Stents With Non-coated Stents
Brief Title: Comparison of Antimicrobial Coated Ureteral Stents With Non-coated Stents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Assisstant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Antimicrobeal ureteral stents
Record Dates: First submitted 2014-10-11; First posted 2014-10-17 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Quality of Life
Keywords: Ureteral stents; Double J stent; Antimicoreal coated stent; USSQ; UTI

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): This arm will include patients with non-coated stents
- Antimicrobeal group (Active Comparator): This arm will include patients with antimicrobeal coated stents
  Interventions: Device: Antimicrobeal coated stents

INTERVENTIONS:
Device: Antimicrobeal coated stents — Patients in the intervention arm will undergo placement of (Silver Sulphdiazine) antimicrobeal coated stents
  Arms: Antimicrobeal group

SUMMARY:
This study will be conducted to compare the efficacy of antimicrobial coated ureteral stent with non-coated stents in prevention of UTI in patients with ureteral stents

DETAILED DESCRIPTION:
The efficacy of antimicrobial coated of ureteral stent with silver sulphadiazine in prevention of UTI in patients with ureteral stents will be studied by comparining the results of urine and stent cultures with patients who had non-coated ureteral stents. The impact of antimicrobeal stent coating on patients' quality of life will be evaluated with comparing the scores of ureteral stent symptom questionnaire between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo ureteral stent placement

Exclusion Criteria:

* Patients allergic to sulpha containing medications
* Ureteral stent insertion for infected hydronephrosis
* Patients who developed septic complications requiring antibiotic treatment after stent placement
* Patients who need bilateral stents
* Patients with chronic kidney disease grade IV and V (GFR <30ml/min)
* Immunocompromised patients as those with malignancy or organ transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of urinary tract infection (UTI) | up to 3 months
  UTI will be diagnosed with urine and stent culture of stent removal

SECONDARY OUTCOMES:
Quality of life | up to 3 months
  The impact of stent coating on quality of life will be assissed with ureteral stent symptom questionnaire (USSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R EL-NAHAS, MD, Study Director — Assistant Professour, urology department, urology and nephrology center, mansoura university
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt